CLINICAL TRIAL: NCT03363828
Title: The Temporo-spatial Dynamics of Genital Tract Microbiota - an Observational Study in IVF-Freeze All Patients Treated With Estradiol
Brief Title: The Temporo-spatial Dynamics of Genital Tract Microbiota
Status: Completed | Type: Observational
Sponsor: Peter Humaidan (Other)
Collaborators: Statens Serum Institut (Other)
Responsible Party: Sponsor-Investigator, Peter Humaidan, Professor, Regionshospitalet Viborg, Skive
Organization: Regionshospitalet Viborg, Skive (Other)
Other Study IDs: 1-10-72-345-15
Record Dates: First submitted 2017-10-29; First posted 2017-12-06 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female | interventions — estradiol, estriol drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Vaginal, cervical and endometrial. Also semen of patients with male partner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal microbiota: Based on qPCR and Next gen sequencing
- Abnormal microbiota: Based on qPCR and Next gen sequencing
  Interventions: Drug: Estrofem

INTERVENTIONS:
Drug: Estrofem — Patients will be asked to obtain self-collected vaginal swabs from the mid-vagina from the beginning of their Estrofem® treatment
  Groups: Abnormal microbiota

SUMMARY:
The investigators aim to examine the endometrium with state of the art sequencing techniques to investigate the endometrial microbiota. The endometrial microbiota has been perceived to be sterile, however, this seems incorrect from recent studies. Thus, the primary outcome is to compare the rate of ascending infection from the semen to the vagina to the endometrium and to investigate which bacteria are capable of inhabiting these environments. Furthermore, cervical mucus will be obtained in order to test for immunological, microbiological and mechanical properties that may be involved in ascending infection. Finally, the study aim to characterize the temporal changes in the vaginal microbiota during estrogenic treatment with Estrofem® or Vivelle Dot (R) for preparation of the endometrium prior to embryo transfer.

ELIGIBILITY:
Inclusion Criteria:

* Patients in IVF Freeze-all/segmentation treatment protocol.
* Written informed consent.

Exclusion Criteria:

* Uterine malformations
* HIV, Hepatitis B or C positivity. HPV CIN 2 or higher. Chlamydia trachomatis positivity.
* Any uncontrolled concomitant disease (e.g. uncontrolled diabetes, uncontrolled hypertension etc.)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile couples attending IVF treatment and referred to a segmentation protocol.
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2021-01-08 (Actual)

PRIMARY OUTCOMES:
Rate of ascending infection/sharing of bacteria in the genital tract | This outcome data is measured at the day of oocyte retrieval.
  Seminal, vaginal, cervical and endometrial samples will be compared at the time of oocyte retrieval.

SECONDARY OUTCOMES:
Next generation sequencing techniques will be used to assess the vaginal microbiota.I.e. measure of relative abundances | Examined longitudinally throughout the segmentation cycle. The estimated time to event is 40 days from oocyte retrieval until frozen embryo transfer following a strict protocol.
  Vaginal microbiota changes throughout the preparation of the endometrium for frozen embryo transfer.
qPCR to assess the vaginal microbiota. I.e. a quantitative measure Copies/mL. | Examined longitudinally throughout the segmentation cycle. The estimated time to event is 40 days from oocyte retrieval until frozen embryo transfer following a strict protocol.
  Vaginal microbiota changes throughout the preparation of the endometrium for frozen embryo transfer.
Number of participants with a Clinical pregnancy | 7-9 weeks after inclusion.
  Tested by clinical pregnancy scan by ultrasound in week 7-9
Number of participants with a Live birth | 36-42 weeks after inclusion
  Tested by self-reported schemes

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - The Fertility Clinic Skive, Skive
  - The Fertility Clinic, Regional Hospital of Skive, Skive

IPD SHARING:
Plan to Share IPD: Yes
Part of PhD project. Data will appear in the thesis and subsequent publications.
Supporting Information: Study Protocol, ICF, CSR